CLINICAL TRIAL: NCT00688116
Title: A Phase 1 Study of the HSP90 Inhibitor, STA-9090, Administered Twice-Weekly in Patients With Solid Tumors
Brief Title: Study of STA-9090, Administered Twice-Weekly in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-01
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumors
Keywords: metastatic cancer; solid tumor; histologically or cytologically confirmed non-hematological malignancy that is metastatic or unresectable; STA-9090; ganetespib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ganetespib (Experimental)
  Interventions: Drug: STA 9090 (ganetespib)

INTERVENTIONS:
Drug: STA 9090 (ganetespib) — This is a dose-escalation study. The first cohort will consist of three patients who will receive 2 mg/m2 of STA 9090 (ganetespib) during a 1-hour infusion 2 times per week (e.g., [Monday, Thursday] or [Tuesday, Friday]) for three consecutive weeks followed by a 1 week dose-free interval. Subsequent cohorts will receive 4, 7, 10, 14, 19, 25, 33, 40 and 48 mg/m2 provided that the previous dose was well tolerated during cycle 1 (week 1 - 4). Further dose increments will be approximately 20% over the previous dose level, until the maximum tolerated dose (MTD) is determined.

SUMMARY:
An open-label dose escalation study of patients with solid tumors treated with STA-9090 (ganetespib)

DETAILED DESCRIPTION:
This is an open-label Phase 1 dose-escalation study in patients with solid tumors treated with STA-9090 (ganetespib) to evaluate for safety, tolerance and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be documented to be refractory or not candidates for current approved therapies. - Must have anECOG status 0-2. - Peripheral neuropathy ?2.
* Must have acceptable organ and marrow function per protocol parameters.
* No clinically significant ventricular arrythmias or ischemia.

Exclusion Criteria:

* Must not be pregnant or breastfeeding. -No chemotherapy or radiation within 3 weeks..
* No previous radiation to >25% of total bone marrow.
* No previous high dose chemotherapy with autologous or allogeniec hematopoietic stem cell transplantation.
* No primary brain tumors or active brain metastases.
* No use of any investigational agents within 4 weeks.
* No treatment with chronic immunosuppressants.
* No uncontrolled, intercurrent illness.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-10; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of STA-9090 (ganetespib) in cancer patients via assessment of dose limiting toxicities and evaluation of Adverse Events in relation to Study Drug. | Cycle 1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA, Los Angeles, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC) - Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan